CLINICAL TRIAL: NCT04873973
Title: Optimized Acute Care for Geriatric Patients Using an Intersectoral Telemedical Cooperation Network - Around the Clock - Technical Performance
Acronym: Optimal@NRW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Collaborators: Optimal@NRW Research Group (Unknown)
Responsible Party: Principal Investigator, Jörg Christian Brokmann, Principal Investigator, RWTH Aachen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-019-2
Record Dates: First submitted 2021-03-31; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Emergencies
Keywords: telemedicine; geriatric; early warning score; acute care; nursing home; emergency department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: Stepped-Wedge-Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in this group are routinely treated.
- Telemedical support (Active Comparator): Participants in this group are routinely treated with additional telemedical support and the use of the early warning system.
  Interventions: Other: Telemedical support

INTERVENTIONS:
Other: Telemedical support — The nursing homes participating in the project will be equipped with telemedical equipment. This will allow teleconsultations to take place when needed. In addition, an early warning system will be introduced and, within the framework of the teleconsultation, a trained medical assistant can be sent to the care facility if necessary, who can carry out medical activities on site under a physician's delegated instructions. In addition, an electronic patient file will be introduced which can be accessed by the telemedicine physician and the general practitioner.
  Arms: Telemedical support

SUMMARY:
Due to "demographic change", the composition of the population in Germany is changing. The consequence of this change is a population that is getting older on average. A key challenge is the appropriate nursing and medical care of older people in senior residences and care facilities. The increasing workload for nursing staff and doctors in the outpatient sector means that timely care for patients, e.g. in the form of GP visits, cannot always be guaranteed in a timely manner. The results are unnecessary or premature hospital admissions as well as ambulance and emergency care interventions, even though in many cases it is not an acute or even life-threatening event. Furthermore, it has been scientifically proven that hospital admissions can increase the risk of patients becoming confused. The aim of this project is to avoid unnecessary hospital admissions and to enable patients to remain in their familiar surroundings as far as this appears medically justifiable. At the same time, the study aims to improve the medical care of nursing home residents through better networking of medical areas, the use of tele-consultations and an early warning system.

DETAILED DESCRIPTION:
The Optimal@NRW project represents a new cross-sectoral approach to the acute care and support of geriatric people in need of care through the implementation of an early warning system and the integration of a telemedical consultation system in 25 nursing homes in the region of Aachen in Germany. The project focuses on restructuring emergency care in nursing homes and improving cooperation between the actors involved (emergency service, emergency department, general practitioners, nursing staff, etc.). Accordingly, a central emergency number of the statutory health insurance funds is to act as a virtual hub for the care of geriatric patients.

The concrete approach of the project is that the participating nursing homes first contact the medical call centre (116 117) in case of a medical problem. The call centre is then responsible for an initial medical assessment and decides whether the respective GP can be called in or whether a teleconsultation with the "virtual digital desk" (i.e. the medical experts from the emergency department of the University Hospital RWTH Aachen) should be carried out. In addition, mobile nursing assistants (NÄPÄ (Z)) will be introduced as part of the project, who can also support the nursing staff and provide services that can be delegated by doctors - especially if the general practitioner is not available at the time.

In addition, a standardised early warning system is to be established in the nursing homes and its benefits evaluated. This will enable potentially dangerous changes in the state of health of nursing home residents to be detected earlier.

The unique and novel development of the technical concept and the interaction between a central electronic patient record, an early warning system and the telemedical equipment plays a decisive role in the success of the project.

ELIGIBILITY:
Inclusion Criteria:

* Resident of one of the participating nursing homes
* At least 18 years old
* Written informed consent
* Consent of the guardian for residents who are not legally able to give consent

Exclusion Criteria:

* Persons placed in an institution by order of an authority or court
* Persons who are in a dependent or employment relationship with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3073 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of non-realized teleconsultations by request | 6 to 15 months depending on the cluster affiliation
  Number of non-realized teleconsultations by request

SECONDARY OUTCOMES:
Number of system crash while running a teleconsultation | 6 to 15 months depending on the cluster affiliation
  Number of system crash while running a teleconsultation
Number of incorrect data transmissions within the overall system | 6 to 15 months depending on the cluster affiliation
  Number of incorrect data transmissions within the overall system
Duration until the realization of a teleconsultation | 6 to 15 months depending on the cluster affiliation
  Duration until the realization of a teleconsultation
Number of causes that lead to system crash | 6 to 15 months depending on the cluster affiliation
  A system crash is defined as a failure of one of the following three components that cannot be recovered within 5 minutes: Audio connection, visual connection, transmission of vital signs.
Data transmission rate requirement | 6 to 15 months depending on the cluster affiliation
  Data transmission rate requirement
Rate of complications of the early warning system in connection with telemedicine | 6 to 15 months depending on the cluster affiliation
  Rate of complications of the early warning system in connection with telemedicine
Performance of the early warning system | 6 to 15 months depending on the cluster affiliation
  - Number of system errors and terminations
Performance of the early warning system | 6 to 15 months depending on the cluster affiliation
  - Number of alarms in the early warning system
Performance of the early warning system | 6 to 15 months depending on the cluster affiliation
  - Number of false alarms
Performance of the early warning system | 6 to 15 months depending on the cluster affiliation
  - time from early warning system alarm to teleconsultation/physician contact
Performance of the early warning system | 6 to 15 months depending on the cluster affiliation
  - consequences of an alarming early warning system
Performance of the teleconsultation equipment | 6 to 15 months depending on the cluster affiliation
  - Number of complications
Performance of the teleconsultation equipment | 6 to 15 months depending on the cluster affiliation
  - Number of disconnection error or failure of components
Performance of the teleconsultation equipment | 6 to 15 months depending on the cluster affiliation
  - consultation extent
Performance of the teleconsultation equipment | 6 to 15 months depending on the cluster affiliation
  - call duration
Performance of the teleconsultation equipment | 6 to 15 months depending on the cluster affiliation
  - devices used

OTHER OUTCOMES:
Satisfaction survey | 24 months
  Questionnaires and interviews to survey satisfaction about the technical equipment in the project
Ethic survey | 24 months
  Questionnaires and interviews to clarify whether the technical equipment is seen as ethically appropriate
Acceptance survey | 24 months
  Questionnaires and interviews to survey acceptance about the technical equipment in the project
Usability survey | 24 months
  Questionnaires and interviews to survey the usability of the technical equipment

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Christian Brokmann, PD Dr. med., Principal Investigator — Uniklinik RWTH Aachen
Locations (1):
- University Hospital RWTH Aachen, Aachen, Germany

REFERENCES:
- [Background] Brown CA, Lilford RJ. The stepped wedge trial design: a systematic review. BMC Med Res Methodol. 2006 Nov 8;6:54. doi: 10.1186/1471-2288-6-54. PMID 17092344
- [Background] Hemming K, Haines TP, Chilton PJ, Girling AJ, Lilford RJ. The stepped wedge cluster randomised trial: rationale, design, analysis, and reporting. BMJ. 2015 Feb 6;350:h391. doi: 10.1136/bmj.h391. No abstract available. PMID 25662947
- [Background] Hoffmann F, Schmiemann G. Influence of age and sex on hospitalization of nursing home residents: A cross-sectional study from Germany. BMC Health Serv Res. 2017 Jan 19;17(1):55. doi: 10.1186/s12913-017-2008-7. PMID 28103927
- [Background] Sundmacher L, Fischbach D, Schuettig W, Naumann C, Augustin U, Faisst C. Which hospitalisations are ambulatory care-sensitive, to what degree, and how could the rates be reduced? Results of a group consensus study in Germany. Health Policy. 2015 Nov;119(11):1415-23. doi: 10.1016/j.healthpol.2015.08.007. Epub 2015 Sep 2. PMID 26428441
- [Background] Vossius C, Selbaek G, Saltyte Benth J, Bergh S. Mortality in nursing home residents: A longitudinal study over three years. PLoS One. 2018 Sep 18;13(9):e0203480. doi: 10.1371/journal.pone.0203480. eCollection 2018. PMID 30226850
- [Background] Bundesärztekammer. Beschlussprotokoll des 121. Deutschen Ärztetages in Erfurt vom 08. bis 11.05.2018, Stand 08.06.2018.
- [Background] Eatock D. Demografischer Ausblick für die Europäische Union 2019.
- [Background] Fehr A, Lange C, Fuchs J, Neuhauser H, Schmitz R. Gesundheitsmonitoring und Gesundheitsindikatoren in Europa. Robert Koch-Institut, Epidemiologie und Gesundheitsberichterstattung; 2017.
- [Background] Jacobs K, Kuhlmey A, Greß S, Klauber J, Schwinger A. Pflege-Report 2018. Berlin, Heidelberg: Springer Berlin Heidelberg; 2018.
- [Background] Sachverständigenrat zur Begutachtung der Entwicklung im Gesundheitswesen. Bedarfsgerechte Steuerung der Gesundheitsversorgung. Gutachten 2018.